CLINICAL TRIAL: NCT01297374
Title: EFFECT OF THREE NON-DRUG INTERVENTION IN TREATMENT OF CHILDREN WITH OVERWEIGHT
Acronym: AMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Claudia Hallal Alves Gazal, Universidade Federal do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCPA100011; HCPA2010 (Other: HCPA)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- dietetic counseling (Experimental)
  Interventions: Behavioral: physical activities, dietician counseling and behavioral changes
- physical activities (Experimental)
  Interventions: Behavioral: physical activities, dietician counseling and behavioral changes
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: physical activities, dietician counseling and behavioral changes

INTERVENTIONS:
Behavioral: physical activities, dietician counseling and behavioral changes — One arm receive an schedule for physical activities. One arm receive a diet prescription. One arm receive general guidance on diet, physical activity and behavioral changes

SUMMARY:
The purpose of this study is to compare the effect of three different non-pharmacological interventions (usually practiced in ambulatory care of Childhood Obesity (AmO), physical activity program (IFSP) and diet therapy adjusted estimate by indirect calorimetry) on the percentage of body fat and basal metabolism of children and Overweight and obesity in the metropolitan region of Porto Alegre (RS).

ELIGIBILITY:
Inclusion Criteria:

* age 8 to 15 years old with overweight (Z-score BMI +1 e +2) and obesity (Z-score BMI > +2)

Exclusion Criteria:

* chronic diseases

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Changes in percentage body fat and basal metabolism after 1 year of randomization | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil